CLINICAL TRIAL: NCT04062292
Title: Investigation of Gait Parameters and Balance in Patients With Obstructive Lung Diseases
Brief Title: Gait Parameters and Balance in Patients With Obstructive Lung Diseases
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Naciye Vardar-Yagli, Associate Professor, Hacettepe University
Other Study IDs: GO 19/665
Record Dates: First submitted 2019-08-15; First posted 2019-08-20 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Gait Disorder, Sensorimotor
Keywords: balance; chronic obstructive diseases
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obstructive lung diseases group: 1. Having been diagnosed with obstructive pulmonary disease,
  2. No acute exacerbation or infection in the past 1 week, Being between the ages of 18 and 65,
- Healthy group: Age and sex matched healthy subjects without orthopedic and chronic diseases

SUMMARY:
In the literature, most of the studies examining the gait characteristics and balance separately or examining the relationship between them are on patients with COPD.

No study examining gait parameters in other obstructive pulmonary patients such as bronchiectasis and asthma was found.A convincing link between gait disturbances and falls in COPD patients is still unknown and further research is needed. Therefore, the purpose of our study; gait parameters and balance in individuals with obstructive pulmonary disease. We will also examine the relationship between gait parameters and extrapulmonary clinical indicators of these individuals.

DETAILED DESCRIPTION:
Patients with COPD call walking as one of the most problematic activities in daily life. Patients with COPD walk less in daily life than their healthy peers. Gait characteristics of extrapulmonary comorbidities that probably affect the musculoskeletal and cardiovascular system vary. The gait assessment gives an idea about the biomechanical factors associated with a reduction in walking distance in COPD patients. In patients with COPD, after the onset of shortness of breath or leg fatigue, a decrease in cadence during walking, shortened stride length, an increase in the time spent in the double support period, an increase in the peak ankle dorsi flexion moment is observed. During gait, there is an increase in balance disorders in the mediolateral direction. In addition, patients with COPD walk on a constant speed treadmill with more stride time and less step width variability. Studies have shown that patients with COPD have increased temporal walking characteristics, decreased step and stride length, and increased walking variability.

In the literature, most of the studies that examine gait characteristics and balance separately or examine the relationship between them are on patients with COPD. No study examining gait parameters in other obstructive pulmonary patients such as bronchiectasis and asthma has been found. A persuasive link between walking disorders and falls in COPD patients is still unknown and further research is needed. This study will contribute to clarifying the mechanisms of why the balance studied in patients with COPD is adversely affected.

ELIGIBILITY:
Inclusion Criteria for Obstructive Lung Diseases

1. Being diagnosed with obstructive lung disease,
2. Have not experienced acute exacerbation or infection in the last 1 week,
3. To be between 18-65 years,
4. Volunteering for research,
5. To be able to walk and cooperate.

Exclusion Criteria for Obstructive Lung Diseases:

1. Use walking aid or be chronic oxygen support
2. To have orthopedic or neuromuscular comorbidities that may affect walking patterns.
3. Having had lung cancer, sarcoidosis, tuberculosis disease or lung surgery.

Inclusion Criteria for Healthy People 1.18-65 years of age, 2. Volunteer to participate in the research, 3. To be able to walk and cooperate.

Exclusion Criteria for Healthy People

1. Having any cardiopulmonary disease,
2. To have an advanced orthopedic disease that may affect functional capacity measurement and gait patterns.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The obstructive lung diseases from every subgroups: COPD, asthma and bronchiectasis patients
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-07-17 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Gait parameters | 01.09.2020-08.07.2021
  Gait parameters will be assessed with Biodex Gait Trainer (Biodex Medical Systems, Shirley, New York) for six minutes.

SECONDARY OUTCOMES:
Functional Balance and Fall Risk | 01.09.2020-08.07.2021
  Timed Up and Go Test
Functional Exercise Capacity | 01.09.2020-08.07.2021
  6 minute walking test with Moxy device on M.Vastus Lateralis
Respiratory Muscle Strength | 01.09.2020-08.07.2021
  Respiratory muscle strength parameters (maximal inspiratory and maximal expiratory pressure) measurement using mouth pressure device
Peripheral Muscle Strength | 01.09.2020-08.07.2021
  Muscle strength of the knee extensors, hip extensors, shoulder abductors, trunk flexors and trunk extensors will be evaluated by hand dynamometer (Lafayette Manual Muscle Tester Model 01165-USA). Jamar Hand Dynamometer (USA) will measure the hand grip force
Cognitive Status | 01.09.2020-08.07.2021
  Mini Mental Test

CONTACTS AND LOCATIONS:
Overall Officials: Naciye Vardar-Yagli, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Naciye Vardar-Yagli, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No